CLINICAL TRIAL: NCT06316206
Title: The Use of Ethinylestradiol/Dienogest in Random Start Rapid Preparation of Endometrium Before Office Hysteroscopic Polypectomies: a Multicenter, Prospective, Randomized Study
Brief Title: The Use of Ethinylestradiol/Dienogest in Random Start Rapid Endometrial Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFIPREP
Record Dates: First submitted 2024-03-07; First posted 2024-03-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Polyp; Endometrial Diseases
Keywords: Hysteroscopy; Endometrial preparation
MeSH Terms: conditions — Uterine Diseases | interventions — Ethinyl Estradiol; dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients with endometrial polyps undergone hysteroscopic polipectomy without endometrial preparation.
- Treatment (Experimental): Patients with endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral Ethinylestradiol/Dienogest 0.03mg/2mg at any time of the menstrual cycle
  Interventions: Drug: Ethinylestradiol/Dienogest 0.03mg/2mg

INTERVENTIONS:
Drug: Ethinylestradiol/Dienogest 0.03mg/2mg — Endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral Ethinylestradiol/Dienogest 0.03mg/2mg at any time of the menstrual cycle
  Arms: Treatment

SUMMARY:
The presence of a thin endometrium plays an important role in enabling the best conditions for hysteroscopic surgery. Recently, for this purpose, many studies have evaluated the effect of preoperative administration of a variety of drugs. We explored the efficacy of random started 14-day administration of Ethinylestradiol/Dienogest, in rapid preparation of endometrium for hysteroscopic polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endometrial polyps.

Exclusion Criteria:

* Patients with other endometrial pathologies.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Quality of endometrial preparation | 14th day of treatment
  Quality of endometrial preparation assessed visually intraoperatively by the surgeon using a visual analog scale from 0 to 5.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Andrea Etrusco, Palermo
  - Marco Monti, Roma

REFERENCES:
- [Derived] Etrusco A, D'Amato A, Agrifoglio V, Chiantera V, Russo G, D'Auge TG, Monti M, Riemma G, Lagana AS, Giannini A. Rapid and random-start endometrial preparation before outpatient hysteroscopic polypectomy in patients of perimenopausal age. Climacteric. 2024 Dec;27(6):561-567. doi: 10.1080/13697137.2024.2404574. Epub 2024 Sep 27. PMID 39329272